CLINICAL TRIAL: NCT04576052
Title: Antibiotic-coated and Uncoated Titanium Nails in Tibia Fractures and Revision Cases Retrospective Cohort Study/ Long-term Clinical Follow-up
Brief Title: Long-term Coated and Non-coated Tibia Nails
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Muenster (Other)
Collaborators: Synthes GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: Protect longterm; DPS-TCMF-2017-042 (Other: Synthes Gmbh)
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Implant Infection
Keywords: fracture associated infection; antibiotic coating; infection prophylaxis; tibia nail; fracture long bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antibiotic-coating: patients who have been treated with an antibiotic-coated nail for tibia-fracture
- non-coated: patients who have been treated with a non-coated nail for tibia fracture

SUMMARY:
For this retrospective cohort study, medical records of patients treated between 2005 to 2019 with the UTN PROtect and/or ETN PROtect for tibia fractures or tibia revision cases will be examined. In comparison to this cohort, patients who received an uncoated tibia nail are examined as well. Demographics, pre-surgical health status, details on fracture type or on revision, treatment decision and surgery details, postoperative reoperation and revision, surgical site infections, time to union, and adverse events will be registered. In a subgroup, additional information including clinical outcomes and patient satisfaction will be assessed by clinical exam. Patients who still carry a nail and feel discomfort at the surgical site or present with a medical condition which demands an imaging will receive an x-ray of the tibia. The xray is not part of the standard study protocol.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective is to assess the proportion of patients who experienced a surgical site infection. Surgical site infection is defined as either deep or superficial. The presence of tibia infection will be defined by the criteria of CDC.

Secondary Objective(s):

* Proportion of patients with reoperation (secondary procedures)
* Bone union (until radiographically healed)
* Proportion of patients with complications / Adverse Events related to implant or surgery
* Only Subgroup: WOMAC-Score, AOFAS, SF36, EQ5D.

Hypothesis and Statistical considerations and estimated enrollment:

We hypothesize that with the use of antibiotic coating implants like the ETN/ UTN-PROtect the risk of implant-associated infections and osteomyelitis is reduced in treatment of Tibia fractures or in cases of revision surgery in the tibia. In a retrospective manner the implanted gentamicin-coated and uncoated tibia nail procedures are evaluated. In the subgroup of patients with a currently implanted gentamicin-coated nail the incidence of surgical site infection and implant-associated infections will be assessed prospectively.

This study is exploratory in nature. Therefore, there is no formal statistical hypothesis and no formal sample size calculation. Approximately 620 tibial shaft fractures are expected to be included in the 12 months enrollment period.

Data will be analyzed with the use of simple summary statistics. Depending on the volume and quality of the collected data, different statistical analyses will be applied. Exploratory analyses will be conducted to investigate relationships between the different treatment options and the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary tibial shaft fracture (fracture type 42 according to the AO/OTA Fracture and Dislocation Classification) treated operatively with an intramedullary nail as Standard of care.
* Signed informed consent, if required by IRB/EC

Exclusion Criteria:

- Prisoner at date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with implantation of a tibial nail to for fracture management or revision surgery
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2020-07-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
infection | 15 years maximum
  Occurrence and time-point of surgical site infection

SECONDARY OUTCOMES:
fracture consolidation | 15 years maximum
  Number of patients with radiographically confirmed bone healing
complications/Adverse Events related to implant or surgery | 15 years maximum
  The occurrence, type, and date of complications/Adverse Events related to implant or surgery
Duration of postoperative immobilization and non-weight bearing | 15 years maximum
  Duration of postoperative immobilization and non-weight bearing as documented in the patient chart

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Raschke, Prof. Dr., Principal Investigator — University Hospital Muenster; Steffen Roßlenbroich, Dr., Principal Investigator — University Hospital Muenster
Locations (1):
- Universtiy Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No